CLINICAL TRIAL: NCT02279758
Title: A PHASE II PILOT STUDY OF METFORMIN TREATMENT IN PATIENTS WITH WELL-DIFFERENTIATED NEUROENDOCRINE TUMORS
Brief Title: A Pilot Study of Metformin Treatment in Patients With Well-differentiated Neuroendocrine Tumors
Acronym: MetNet
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Instituto do Cancer do Estado de São Paulo (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NP 515/2014
Record Dates: First submitted 2014-07-07; First posted 2014-10-31 (Estimated); Last update posted 2014-10-31 (Estimated); Status verified 2014-10

CONDITIONS: Well-differentiated Neuroendocrine Tumors
Keywords: Neuroendocrine Tumors; The Mammalian Target of Rapamycin (mTOR); metformin
MeSH Terms: conditions — Neuroendocrine Tumors | interventions — Metformin

ARMS (1):
- METFORMIN (Experimental): 850mg of metformin every 12 hours.
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin

SUMMARY:
Neuroendocrine tumors are rare but recent data showed a relevant increase in its incidence. The Mammalian Target of Rapamycin (mTOR), one of most important area of research, has demonstrated be a therapeutic target in these tumors. The metformin has demonstrate in preclinical studies having an antineoplastic action by inhibiting the mTOR pathway, and may be an alternative treatment for this disease.

Eligible patients for this study should have metastatic gastroenteropancreatic neuroendocrine tumors well differentiated (grade 1 or grade 2) and will be treated with metformin 850 mg every 12 hours, and each cycle will consist of 30 days. After 180 days of treatment the efficacy of metformin under the control of disease progression will be evaluated. As a secondary outcome the investigator will check the patient adherence to the treatment, the control of patient symptoms with functioning neuroendocrine tumor, and disease free survival. Also will be performed an analysis of immunohistochemical expression of mTOR pathway proteins of these patients.

ELIGIBILITY:
Inclusion Criteria:

* Metastatic well-differentiated neuroendocrine tumor grade 1 or 2 with histological confirmation;
* Performance status according to Eastern Cooperative Oncology Group (ECOG) 0 to 2;
* Able to take pills;
* Age ≥ 16 years;
* Ability to Provide Written Informed Consent;
* Adequate organ function;

Exclusion Criteria:

* Patient with out of control severe hormonal syndrome;
* Diabetic patients under metformin treatment, or those who have received treatment with metformin within 3 months;
* Patient with hypersensitivity to biguanides, kidney or liver failure, or other conditions that predispose to lactic acidosis;
* History of severe clinical or psychiatric illness, that would prevent participation in the study by clinical judgment;
* Patients who participate in other protocol with experimental drugs;
* Patients under any kind of active infection;
* Patients who have received chemotherapy within 3 weeks;
* Patients pregnant or lactating;
* Diabetic patients who require higher dose of metformin 850mg x 2 daily;

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2014-03; Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Disease free survival | After 180 days of treatment.

SECONDARY OUTCOMES:
Number of Participants with Adverse Events Related to Metformin Measured of Safety and Tolerability | Assessments will be performed until 180 days after treatment initiation
  Clinical evaluation of metformin related toxicity will be assessed at each medical visit (once a month).
Clinical benefit | Assessments will be performed until 180 days after treatment initiation.
  Clinical benefit will be measured using CTCAE version 4.03 for analysis of adverse events presented by patients.
Biochemical response | Assessment will be performed at day 90 and 180 of treatment.
  Biochemical response defined by tumor markers.
Evaluation of patient's glycemic profile | Assessment will be performed at day 90 and day 180 of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: João Glasberg, MD, Principal Investigator — Instituto do Cancer do Estado de São Paulo
Locations (1):
- Instituto do Cancer do Estado de São Paulo, São Paulo, São Paulo, Brazil